CLINICAL TRIAL: NCT04585503
Title: Feasibility Study of Cortical Recording Depolarizations in Brain-injured Patients, and Their Use as Biomarkers of New Lesions.
Acronym: SD-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0615
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Brain Lesion; Head Trauma; Subarachnoid Hemorrhage
Keywords: subdural or intra cortical implanted electrodes; CNS monitor; brain lesions
MeSH Terms: conditions — Craniocerebral Trauma; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Central nervous system monitoring (Experimental): Each 20 patients will be implanted with subdural or intra cortical electrodes
  Interventions: Device: Electrode implantation

INTERVENTIONS:
Device: Electrode implantation — The intervention consist in implanting 6 electrodes in subdural or intra cortical position and monitor the central nervous system activity. This monitoring will be additional to the usual monitoring.

SUMMARY:
The progression of brain lesions after severe head trauma or subarachnoid hemorrhage results from extra cranial aggression which is well controlled in intensive care and intracranial aggression which is less well known and therefore less well managed. The detection of events that can generate new lesions from intracranial monitoring is limited and late once the lesions are irreversible. Invasive cortical depolarizations (SD) can be observed using cortical electrodes and an acquisition system having access to the usually filtered DC signal (0 to 1 Hz). SD are observed at the onset of a new attack of the cortex and spread widely away from the site of aggression. During their propagation, SD generate a significant metabolic demand, and can cause ischemic injury, particularly after meningeal or post-traumatic hemorrhage. SDs are therefore both a marker of new lesion and a mechanism of progression of primary lesions. Yet this type of monitoring is only performed in some expert centers around the world. The analysis of the feasibility and safety of the placement of cortical electrodes in this indication is therefore an essential step to study the clinical benefit of individualized management on the basis of this monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 year old
* Patients admitted in neurological reanimation unit for brain lesions after severe head trauma or subarachnoid hemorrhage and requesting a intracranial monitoring or a surgery (evacuation of a hematoma, treatment of an aneurysm, external ventricular bypass).
* Patients affiliated to a social security system
* Patient having been informed and having signed the Consent form OR Close to the patient who has been informed and signed the Consent form OR third party certificate then close consent for further study.

Exclusion Criteria:

* Patient with scalp acute infection
* Pregnant or nursing women
* Contre-indication to intracranial surgery
* Patient with not corrected coagulation disorder
* Patient treated with NSAIDS
* Patient treated with under platelet antiaggregants
* Patient under legal protection, guardianship, curators
* patients under legal protection
* Patient participating in a study who may interfere with this study.
* people under duress psychiatric care,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of Invasive cortical depolarization (SD) recorded in a non-expert center with subdural or intra cortical implanted electrode and central nervous system monitoring. | 18 months
  The feasibility of the study will be objectivized by the availability of a signal of sufficient quality to be exploited, with or without SD: namely a signal without artifact on more than 30% of the recording period on at least 3 electrodes on 6 for at least 12h. The signal analysis should, at least twice a day, allow intervening with the patient if necessary.

SECONDARY OUTCOMES:
Evaluation of electrode implantation safety | during implantation procedure
  Safety will be evaluated recording severe and non-severe adverse events during implantation procedure.
Evaluation of electrode implantation safety | during monitoring, maximum 15 days
  Safety will be evaluated recording severe and non-severe adverse events during monitoring
Evaluation of electrode implantation safety. | during electrode extraction
  Safety will be evaluated recording severe and non-severe adverse events during electrode extraction.
Evaluation of temporality between Invasive cortical depolarization and intracranial hypertension. | during monitoring, maximum 15 days
  proportion of patient with Invasive cortical depolarization before, during and after intracranial hypertension.
Evaluation of temporality between Invasive cortical depolarization and oxygen in tissue decreasing pressure | during monitoring, maximum 15 days
  proportion of patient with Invasive cortical depolarization before during and after oxygen in tissue decreasing.
Evaluation of temporality between Invasive cortical depolarization and detection of a vasospasm | during monitoring, maximum 15 days
  proportion of patient with Invasive cortical depolarization before during and after detection of a vasospasm.
Evaluation of temporality between Invasive cortical depolarizations and EEG change of rhythm. | during monitoring, maximum 15 days
  proportion of patient with Invasive cortical depolarization before, during and after EEG change of rhythm.
Evaluation of temporality between Invasive cortical depolarization and detection of a new cerebral lesion. | during monitoring, maximum 15 days
  proportion of patient with Invasive cortical depolarization before, during and after detection of a new cerebral lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie réanimation Groupement hospitalier Est, hôpital Pierre Wertheimer, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghibaudo V, Bado J, Garcia S, Berthiller J, Rithzenthaler T, Gobert F, Bapteste L, Carrillon R, Bodonian C, Dailler F, Haegelen C, Dumot C, Rheims S, Berhouma M, Balanca B. Lessons to Learn from Multimodal Neuromonitoring of Brain Death with Electrophysiological Markers of Cortical and Subcortical Loss of Functions. Neurocrit Care. 2024 Dec;41(3):1110-1114. doi: 10.1007/s12028-024-02049-4. Epub 2024 Jul 9. No abstract available. PMID 38982002
- [Derived] Balanca B, Ghibaudo V, Bado J, Berthiller J, Ritzenthaler T, Gobert F, Bapteste L, Carrillon R, Bodonian C, Contard F, Percevault G, Marinesco S, Dreier JP, Woitzik J, Haegelen C, Rheims S, Dumot C, Dailler F, Berhouma M. Feasibility and safety of electrocorticography monitoring after acute brain injury to detect cortical spreading depolarisation, a prospective observational study in a neurological intensive care unit. Anaesth Crit Care Pain Med. 2025 Nov 13:101669. doi: 10.1016/j.accpm.2025.101669. Online ahead of print. PMID 41241268